CLINICAL TRIAL: NCT01390662
Title: Phase 4 Study of Vitamin D3 Supplementation for Outcomes in Patients With Unipolar Depression
Brief Title: Can Vitamin D3 Supplementation Affect Treatment Outcomes in Patients With Depression
Acronym: D3-vit-dep
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Syddanmark (Other)
Responsible Party: Connie Thuroee Nielsen, consultant,PhD, Mental Health Services Esbjerg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26992; 2010-023531-42 (EudraCT Number)
Record Dates: First submitted 2011-07-05; First posted 2011-07-11 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2011-07

CONDITIONS: Depression
Keywords: serum 25-hydroxyvitamin d,vitamin D supplement, depression,; parathyroid hormone
MeSH Terms: conditions — Depression | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Active Comparator): one tablet of vitamin D3 (70µg) per day for 24 weeks.
  Interventions: Dietary Supplement: Vitamin D3
- placebo (Placebo Comparator): one tablet of sugar pill per day for 24 weeks.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — one tablet of vitamin D3 70 µg pr. day, for 24 weeks.
  Arms: Vitamin D3
Dietary Supplement: placebo — one tablet of sugar pill pr. day, for 24 weeks.
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate whether patients with depression should be offered vitamin D supplements, or it has no significance in relation to treatment outcomes.

DETAILED DESCRIPTION:
Vitamin D3 is produced in the skin after exposure to ultraviolet B light from the sun. Vitamin D3 is metabolised sequential in the liver into 25-hydroxy-vitamin D [25(OH)D], which is the storage form of vitamin D in the body, and then in the kidney into the steroid hormone, 1a,25-dihydroxyvitamin 1a,25-dihydroxyvitamin D [1,25(OH)2D].

At higher latitudes ultraviolet B light is stopped by the atmosphere during winter season. Half of Danes have low levels of [25(OH)D] in the blood and especially in the early spring months the levels of [25(OH)D] are low. In addition, Vitamin D3 is absorbed through the gut from vitamin D-rich food sources. But several studies show that it is not possible through a recommended diet, which consists of 300 g of fish per week to consume adequate amounts of vitamin D3.

New research suggests link between vitamin D3 and brain function.In the Central Nervous System (CNS) there are specific nuclear receptors for 1,25(OH)2D (VDR) and the enzymes necessary for the hydroxylation of 25(OH)D to 1,25(OH)2D are also present in CNS.

In clinical studies, low serum levels of 25(OH)D, have been associated with reduced cognitive function, anxiety and depression.

The objective of this randomized clinical trial is to investigate whether patients with depression should be offered vitamin D3 supplements, or it has no significance in relation to treatment outcomes.

The study is carried out in Mental Health Services in the Region of Southern Denmark for 24 weeks and offered to patients being treated for depression (treatment as usual) plus 70μg vitamin D3 or placebo.

ELIGIBILITY:
Inclusion Criteria

* clinical diagnosis unipolar depression

Exclusion Criteria:

* clinical diagnosis sarcoidoses
* tuberculosis
* bipolar affective disorder
* schizophrenia
* hypercalcemia
* hyperphosphatemia
* electroconvulsive treatment for the last 6 months
* primary diagnosis addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-05 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton 17 item scale (Hamilton-17) | 24 weeks
  Change from baseline in Hamilton-17 at week 24

SECONDARY OUTCOMES:
WHO-Five Well-being Index (WHO-5) | 24 weeks
  Change from baseline in WHO-five at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Connie T Nielsen, PhD, Study Chair — Mental Health Services Esbjerg; Erik Dahl, MD, Principal Investigator — Mental Health Services Svendborg; Tomas toft, PhD, Principal Investigator — Mental Health Services Odense
Locations (3):
- Denmark (3):
  - Mental Health Services Esbjerg, Esbjerg
  - Mental Health Services, Odense, Odense
  - Mental Health Services Svendborg, Svendborg

REFERENCES:
- [Derived] Hansen JP, Pareek M, Hvolby A, Schmedes A, Toft T, Dahl E, Nielsen CT. Vitamin D3 supplementation and treatment outcomes in patients with depression (D3-vit-dep). BMC Res Notes. 2019 Apr 3;12(1):203. doi: 10.1186/s13104-019-4218-z. PMID 30944021